CLINICAL TRIAL: NCT03677882
Title: A Randomized Pilot Study of a Brief Mind-Body Bridging Intervention for Suicidal Ideation
Brief Title: A Brief Mind-Body Bridging Intervention for Suicidal Ideation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We experienced recruitment difficulties, and the focus of the department has changed.
Sponsor: VA Salt Lake City Health Care System (U.S. Federal Agency)
Collaborators: Mind Body Bridging Charity (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VASaltLakeCity
Record Dates: First submitted 2018-09-10; First posted 2018-09-19 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Suicidal Ideation; Mind Body Bridging
Keywords: mind body bridging; mindfulness; suicidal ideation; suicide related behaviors
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (TAU) (No Intervention): Participants assigned to Treatment As Usual (TAU) will receive the normal standard of care treatment from the Suicide Prevention Team and the Mental Health Service which may include individual therapy, group therapy, and/or medication therapy, all as decided by the individual and his/her doctor. Treatment as usual also includes monitoring by the Suicide Prevention Team.
- Treatment As Usual with Mind-Body Bridging (TAU + MBB) (Experimental): Participants assigned to TAU + MBB will will receive treatment from the Suicide Prevention Team and the Mental Health Service, AND will be asked to participate in consisting of three to eight 60-minute sessions that will occur consecutively. Each group will be led by a trained MBB facilitator. Participants will receive a workbook at the beginning of the training that contains an explanation of all the major concepts involved in Mind Body Bridging. The workbook has homework assignments to be completed daily between group sessions.
  Interventions: Behavioral: Mind Body Bridging Group Session

INTERVENTIONS:
Behavioral: Mind Body Bridging Group Session — Participants assigned to TAU + MBB will will receive treatment from the Suicide Prevention Team and the Mental Health Service, AND will be asked to participate in consisting of three to eight 60-minute sessions that will occur consecutively. Each group will be led by a trained MBB facilitator. Participants will receive a workbook at the beginning of the training that contains an explanation of all the major concepts involved in Mind Body Bridging. The workbook has homework assignments to be completed daily between group sessions.
  Arms: Treatment As Usual with Mind-Body Bridging (TAU + MBB)

SUMMARY:
The aim of this study is to determine whether a Brief Mind-Body Bridging Intervention for Suicidal Ideation (MBB-SI) will result in short or longer-term reduction of psychological factors associated with suicidal ideation (SI) and/or suicide-related behaviors (SRB's) compared to Treatment as Usual (TAU).

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be Veterans aged 18-80 admitted to Substance Abuse Residential Rehabilitation Treatment Program (SARRTP) with addictive disorders and/or co-occurring psychiatric disorder with suicide risk factors.

Exclusion Criteria:

* None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Change in frequency and/or intensity of suicidal ideation | Weekly during the intervention, one-month post-intervention, three months post-intervention, six months post-intervention
  Determine if there is a significant difference in the frequency and/or intensity of suicidal ideation, as measured by the Beck Scale for Suicide Ideation (BSS) among the MBB-SI + TAU cohort compared to the TAU. We will use the total BSS score, ranging from 0 to 38. Increased scores reflect greater suicide risk.

CONTACTS AND LOCATIONS:
Overall Officials: William Marchand, MD, Principal Investigator — VA Salt Lake City HCS
Locations (1):
- George E. Wahlen Department of Veterans Affairs Medical Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No